CLINICAL TRIAL: NCT04973462
Title: Evaluation of The Efficacy of Triazavirin Versus Oseltamivir in Egyptian Patients Infected With Coronavirus Disease 2019 (COVID-19)
Brief Title: Evaluation of The Efficacy of Triazavirin Versus Oseltamivir in Egyptian Patients Infected With COVID-19
Acronym: COVID-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amal A. Elkholy, Principal Investigator Dr., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Antiviral therapy in COVID-19
Record Dates: First submitted 2021-07-03; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — riamilovir; Oseltamivir

STUDY DESIGN:
Intervention Model Description: Simple Randomization Parallel Double Blinded.
Who Masked: Participant, Care Provider
Masking Description: To ensure blindness one placebo capsule will be added to group B.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triazavirin group (Active Comparator): Patients will take the standard treatment COVID-19 + Triazavirin 250mg three times daily for 7 days]
  Interventions: Drug: standard treatment COVID-19 + Triazavirin
- Oseltamivir group (Active Comparator): Patients will take the standard treatment COVID-19 + Oseltamivir 75 mg twice daily for 7 days]
  Interventions: Drug: standard treatment COVID-19 + Triazavirin

INTERVENTIONS:
Drug: standard treatment COVID-19 + Triazavirin — to evaluate the efficacy and safety (side effects and / or adverse effects) of Triazavirin and Oseltamivir as treatment of Coronavirus Disease 2019
  Other Names: standard treatment COVID-19 + Oseltamivir

SUMMARY:
The aim of this study is to evaluate the efficacy and safety (side effects and / or adverse effects) of Triazavirin and Oseltamivir as treatment of Coronavirus Disease 2019 in Egyptian patients in military hospitals.

DETAILED DESCRIPTION:
In December 2019, a series of pneumonia cases of unknown cause emerged, followed by a rapidly spread due to strong human-to-human transmission in china. Based on the clinical presentation, the pneumonia was determined to be a viral infection; the virus was initially named the 2019 novel coronavirus (2019-nCoV) and then, formally, severe acute respiratory syndrome coronavirus2 (SARS-CoV-2). Most districts have reported zero increase of coronavirus disease 2019 (COVID-19) cases since March 2020. As of 11 March 2020, a total of 80 955 laboratory-confirmed cases had been documented in China.

The World Health Organization (WHO) declared COVID-19 to be a public health emergency of international concern on 30 January 2020. The mortality rate was found to be 3.9% according to the data at that time. Given the human-to-human transmission and high infectivity of the disease, COVID-19 has been rapidly spreading in Republic of Korea, Iran, Italy, the United States, and Europe. A number of studies and reports have identified a median incubation period of 4 d and have determined that the top four symptoms include fever, cough, shortness of breath, and chest tightness/pain.

The most unfortunate fact is that there have been no effective therapies for preventing and treating COVID-19 to date. Although Remdesivir and Hydroxychloroquine have been found to be effective in inhibiting SARS-CoV-2, the data obtained thus far are primarily from in vitro studies, but their effectiveness in vivo still questionable. Interferon, Lopinavir/ritonavir, Arbidol, Ribavirin, and the therapeutic application of plasma antibodies have also been recommended as alternatives for the treatment of patients with COVID-19; however, the efficacy and safety of these drugs remain to be verified in patients, and their applications are yet to be validated by scientifically sound randomized clinical trials (RCTs).

Triazavirin (TZV), a new antiviral drug, has been on the market in Russia since 2015. It is a synthetic compound analogue to the purine nucleoside bases. The principle mode of action of TZV is inhibiting the synthesis of viral RNA and preventing the replication of genomic fragments. Because of its multiple-target mechanism of action, TZV has a wide spectrum of antiviral activity against RNA-containing viruses, including influenza A virus (H5N1, etc.), influenza B virus, tick-borne encephalitis, and Forest-Spring encephalitis, both in vitro and in animal models in vivo.

Oseltamivir is a first-line antiviral drug, especially in primary hospitals of military medical hospitals. During the ongoing outbreak of coronavirus disease 2019 (COVID-19), most patients with COVID-19 who are symptomatic have used Oseltamivir. Considering its popular and important role as an antiviral drug, it is necessary to evaluate oseltamivir in the treatment of COVID-19 . Oseltamivir inhibits the neuraminidase enzyme, which is expressed on the viral surface. The enzyme promotes release of virus from infected cells and facilitates viral movement within the respiratory tract. In the presence of neuraminidase inhibitors, virions stay attached to the membrane of infected cells and are also entrapped in respiratory secretions.

ELIGIBILITY:
Inclusion Criteria:

1. Adults from 18 to 60 years old who signed informed consent;
2. Laboratory confirmed SARS-CoV-2 infection by real-time RT-PCR.
3. Chest computed tomography (CT) imaging-confirmed lung damage, including multiple small plaques and stromal changes in the lungs, which are obvious in the outer lung, or multiple ground-glass shadows and infiltration shadows in both lungs, although these changes might not be present in mild patients.
4. Patients with history of fever (axillary temperature more than 37°С) or respiratory symptoms.

Exclusion Criteria:

1. Patients who are unsuitable or who cannot participate safely in the study, as judged by the principal investigator (PI).
2. Patients with serious liver disease (increase of liver transaminases enzymes).
3. Patients with severe renal impairment (denoted by increase serum urea & serum creatinine) or continuous renal replacement therapy, hemodialysis, or peritoneal dialysis.
4. Patients with severe anemia.
5. Women with a positive pregnancy test, ongoing pregnancy, or who are breastfeeding.
6. Patients with a history of allergy to medications or its metabolic components.
7. Patients who have not signed informed consent.
8. Patients participating in other clinical trials for COVID-19 within 30 days prior to screening.
9. Patients participating in other clinical research in the past three months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Physicians Global Assessment to measure the baseline COVID-19 signs and symptoms | baseline
  1. Temperature response (axillary temperature more than 37°С)
  2. Fever response (axillary temperature more than 37.8°С)
  3. General intoxication symptoms (e.g. headache, myalgia, eyebulb pain)
  4. Catarrhal symptoms (e.g.sore throat, cough).

SECONDARY OUTCOMES:
Time to recovery | 7 days
  (temperature ≤37.0°С, no intoxication symptoms) depending on time of therapy initiation (infection day 1 or 2) in the two groups.
Incidence of re-detection of viral RNA using PCR | 7 days
  (% of patients with positive PCR)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 month
  * Computed Tomography (CT) chest
  * PCR (Polymerase chain reaction)
  * CBC (complete blood count)
  * Serum Ferritin in ug/L
  * Liver & kidney functions
  * Cardiac troponin in ng/L
  * Coagulation profile (INR-PT-PTT in minutes)
  * Blood glucose level in mg/dL
  * Erythrocyte Sedimentation Rate (ESR) in mm/hr
  * C-Reactive Protein (CRP) mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa A Sabri, professor, Study Chair — Department of Clinical Pharmacy
Locations (1):
- Fever Hospital of the Egyptian Armed Forces, Cairo, Egypt

REFERENCES:
- [Background] Chen S, Yang J, Yang W, Wang C, Barnighausen T. COVID-19 control in China during mass population movements at New Year. Lancet. 2020 Mar 7;395(10226):764-766. doi: 10.1016/S0140-6736(20)30421-9. Epub 2020 Feb 24. No abstract available. PMID 32105609
- [Background] Zhang W, Du RH, Li B, Zheng XS, Yang XL, Hu B, Wang YY, Xiao GF, Yan B, Shi ZL, Zhou P. Molecular and serological investigation of 2019-nCoV infected patients: implication of multiple shedding routes. Emerg Microbes Infect. 2020 Feb 17;9(1):386-389. doi: 10.1080/22221751.2020.1729071. eCollection 2020. PMID 32065057
- [Background] Sethi BA, Sethi A, Ali S, Aamir HS. Impact of Coronavirus disease (COVID-19) pandemic on health professionals. Pak J Med Sci. 2020 May;36(COVID19-S4):S6-S11. doi: 10.12669/pjms.36.COVID19-S4.2779. PMID 32582306
- [Background] Lim J, Jeon S, Shin HY, Kim MJ, Seong YM, Lee WJ, Choe KW, Kang YM, Lee B, Park SJ. Case of the Index Patient Who Caused Tertiary Transmission of COVID-19 Infection in Korea: the Application of Lopinavir/Ritonavir for the Treatment of COVID-19 Infected Pneumonia Monitored by Quantitative RT-PCR. J Korean Med Sci. 2020 Feb 17;35(6):e79. doi: 10.3346/jkms.2020.35.e79. PMID 32056407
- [Derived] Mohamed Elmenshawy SS, Ahmed Abdelsalam MF, El Nagdy TR, Salam Elgohary MA, Sabri NA, El-Kholy A. Evaluation of the efficacy of triazavirin versus oseltamivir in management of COVID-19. Future Sci OA. 2024 Dec 31;10(1):2418798. doi: 10.1080/20565623.2024.2418798. Epub 2024 Nov 14. PMID 39539144